CLINICAL TRIAL: NCT05341713
Title: Epileptic Seizure in Epilepsy Patients After First-dose Inactivated SARS-CoV-2 Vaccination: a Self-controlled Case Series Study
Brief Title: Epileptic Seizure in Epilepsy Patients After SARS-CoV-2 Vaccination
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Liu Yonghong, Professor, Xijing Hospital
Other Study IDs: KY20222046-C-1
Record Dates: First submitted 2022-04-16; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Epileptic Seizures Related to Drugs; SARS-CoV-2 Acute Respiratory Disease; Vaccine Adverse Reaction
Keywords: epilepsy patient; risk of seizure; SARS-Cov-2 vaccine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: inactive SARS-Cov-2 vaccine — We included epilepsy patients who were vaccinated with inactive SARS-CoV-2 vaccines

SUMMARY:
Background and Objectives: Seizure attack is one of adverse effects of vaccination in epileptic patients, the risk of which after severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) inoculation was elucidated in the present study.

Methods: A self-controlled case series study was designed to examine the association between vaccination and epileptic seizure. A total of 240 epilepsy patients were included who were vaccinated with inactive SARS-CoV-2 vaccines (Sinovac Life Sciences and Lanzhou Institute of Biological Products) and admitted to outpatient clinics from July 2021 to December 2021. Poisson analysis was performed to estimate the relative incidence rate of epileptic seizure in risk periods (day 1-7, 8-21 and 1-21 after first-dose vaccination) compared to basal level in control period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants
* Have a diagnosis of epilepsy by the end of the study
* Have received at least one dose of inactive SARS-Cov-2 vaccine (Sinovac Life Sciences and Sinopharm Group)

Exclusion Criteria:

* Non-epilepsy patients vaccinated with inactive SARS-Cov-2 vaccine
* Epilepsy patients administrated with non-inactive vaccine
* Unvaccinated epilepsy patients

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We retrospectively enrolled epilepsy patients visiting outpatient clinics of the above two centers from July 2021 to December 2021, who took inactivated vaccines from Sinovac Life Sciences and Sinopharm Group (China). The study included both adults and children aged above 3 years. All the patients were diagnosed with epilepsy according to the International League Against Epilepsy (ILAE) Commission 90 days before till 21 days after the first dose of vaccine. Demographics, clinical manifestations and vaccination records were collected.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Risk of epileptic seizures within 21 days after first-dose vaccination with inactive SARS-CoV-2 vaccine in epilepsy patients | from 90 days before until 21 days after the first dose of vaccine
  Overall relative incidence of epileptic seizures in risk periods compared to control period.
Risk of epileptic seizures in epilepsy patients of different subgroups | from 90 days before until 21 days after the first dose of vaccine
  The associations of sex, age or medication status with the relative incidence in risk periods

CONTACTS AND LOCATIONS:
Overall Officials: Gengyao Hu, doctor, Principal Investigator — Air Force Military Medical University, China; Ze Chen, master, Principal Investigator — Air Force Military Medical University, China; Kejian Wu, doctor, Principal Investigator — Air Force Military Medical University, China; Yuanhang Pan, master, Principal Investigator — Air Force Military Medical University, China; Xia Li, master, Principal Investigator — Xian Children's Hospital; Junxiang Bao, doctor, Study Director — Air Force Military Medical University, China; Yonghong Liu, doctor, Study Chair — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Frontera JA, Sabadia S, Lalchan R, Fang T, Flusty B, Millar-Vernetti P, Snyder T, Berger S, Yang D, Granger A, Morgan N, Patel P, Gutman J, Melmed K, Agarwal S, Bokhari M, Andino A, Valdes E, Omari M, Kvernland A, Lillemoe K, Chou SH, McNett M, Helbok R, Mainali S, Fink EL, Robertson C, Schober M, Suarez JI, Ziai W, Menon D, Friedman D, Friedman D, Holmes M, Huang J, Thawani S, Howard J, Abou-Fayssal N, Krieger P, Lewis A, Lord AS, Zhou T, Kahn DE, Czeisler BM, Torres J, Yaghi S, Ishida K, Scher E, de Havenon A, Placantonakis D, Liu M, Wisniewski T, Troxel AB, Balcer L, Galetta S. A Prospective Study of Neurologic Disorders in Hospitalized Patients With COVID-19 in New York City. Neurology. 2021 Jan 26;96(4):e575-e586. doi: 10.1212/WNL.0000000000010979. Epub 2020 Oct 5. PMID 33020166
- [Background] Cabezudo-Garcia P, Ciano-Petersen NL, Mena-Vazquez N, Pons-Pons G, Castro-Sanchez MV, Serrano-Castro PJ. Incidence and case fatality rate of COVID-19 in patients with active epilepsy. Neurology. 2020 Sep 8;95(10):e1417-e1425. doi: 10.1212/WNL.0000000000010033. Epub 2020 Jun 17. PMID 32554773
- [Background] Frontera JA, Tamborska AA, Doheim MF, Garcia-Azorin D, Gezegen H, Guekht A, Yusof Khan AHK, Santacatterina M, Sejvar J, Thakur KT, Westenberg E, Winkler AS, Beghi E; contributors from the Global COVID-19 Neuro Research Coalition. Neurological Events Reported after COVID-19 Vaccines: An Analysis of VAERS. Ann Neurol. 2022 Mar 2;91(6):756-71. doi: 10.1002/ana.26339. Online ahead of print. PMID 35233819
- [Background] Massoud F, Ahmad SF, Hassan AM, Alexander KJ, Al-Hashel J, Arabi M. Safety and tolerability of the novel 2019 coronavirus disease (COVID-19) vaccines among people with epilepsy (PwE): A cross-sectional study. Seizure. 2021 Nov;92:2-9. doi: 10.1016/j.seizure.2021.08.001. Epub 2021 Aug 6. PMID 34391030
- [Background] Arnheim-Dahlstrom L, Hallgren J, Weibull CE, Sparen P. Risk of presentation to hospital with epileptic seizures after vaccination with monovalent AS03 adjuvanted pandemic A/H1N1 2009 influenza vaccine (Pandemrix): self controlled case series study. BMJ. 2012 Dec 18;345:e7594. doi: 10.1136/bmj.e7594. PMID 23274350